CLINICAL TRIAL: NCT07305337
Title: The Impact of Artificial Intelligence-Assisted Health Education on Patients' Intention to Participate in Clinical Trials: A Cluster-Randomised Controlled Trial
Brief Title: Randomised Controlled Trial of Artificial Intelligence-assisted Health Education
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Fuling Zhou, Dean, School of Nursing, Wuhan University; Tenured Full Professor, Director of Department of Hematology, zhongnan Hospital,Wuhan University, Zhongnan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0603
Record Dates: First submitted 2025-06-03; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Leukaemia; Multiple Myeloma (MM), Lymphoma, Large B-Cell, Diffuse (DLBCL), Lymphoma; Lymphoma
Keywords: Leukaemia; Multiple Myeloma; Lymphoma; health education; artificial intelligence
MeSH Terms: conditions — Leukemia; Multiple Myeloma; Lymphoma; Health Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial Intelligence Health Education (Experimental): In addition to receiving standard health education, participants underwent clinical trial-specific education delivered via an AI robot. This educational content was designed around fundamental concepts of clinical trials, implementation procedures, clarification of common misconceptions, ethical safeguards, and potential benefits of participation. Its aim was to enhance patients' overall understanding of clinical trials and willingness to participate. The AI robot featured voice interaction capabilities and integrated text-image displays with video materials to enhance the interactivity and comprehensibility of information delivery.
  Interventions: Device: Artificial Intelligence Health Education
- Artificial health education (Active Comparator): Received only routine health education delivered by departmental healthcare staff, covering fundamental disease knowledge, treatment protocols, nursing management, and discharge instructions. This education forms part of the hospital's standard clinical practice and typically does not systematically incorporate content related to clinical trials or dedicated educational modules.
  Interventions: Other: Artificial health education

INTERVENTIONS:
Device: Artificial Intelligence Health Education — In addition to receiving standard health education, participants underwent clinical trial-specific education delivered via an AI robot. This educational content was designed around fundamental concepts of clinical trials, implementation procedures, clarification of common misconceptions, ethical safeguards, and potential benefits of participation. Its aim was to enhance patients' overall understanding of clinical trials and willingness to participate. The AI robot featured voice interaction capabilities and integrated text-image displays with video materials to enhance the interactivity and comprehensibility of information delivery.
  Arms: Artificial Intelligence Health Education
Other: Artificial health education — Received only routine health education delivered by departmental healthcare staff, covering fundamental disease knowledge, treatment protocols, nursing management, and discharge instructions. This education forms part of the hospital's standard clinical practice and typically does not systematically incorporate content related to clinical trials or dedicated educational modules.
  Arms: Artificial health education

SUMMARY:
With the rapid advancement of biopharmaceutical technology, clinical trials have become the crucial bridge connecting new drugs from the laboratory to clinical application. Despite the increasing number of clinical trial projects being conducted, nearly all such projects face the common challenge of recruitment difficulties. Subject recruitment constitutes a pivotal stage in clinical trials; the ability to recruit a sufficient number of subjects meeting the trial requirements significantly impacts trial quality and also serves as a key factor influencing trial progress. Hematologic cancers constitute a highly heterogeneous group of malignant diseases originating in the haematopoietic organs and primarily affecting the haematopoietic system. They encompass acute and chronic leukaemias, malignant lymphomas, multiple myeloma, myelodysplastic syndromes, and related disorders. For patients facing treatment decisions, clinical trials represent not only a vital avenue for accessing cutting-edge therapies but also impose heightened demands on their capacity for informed decision-making. Conversational artificial intelligence (AI) based on large language models is rapidly advancing in health education and public health communication. Medical chatbots offer scalable and personalised advantages in delivering health information, promoting behavioural change, and enhancing patient engagement, providing a viable pathway for improving trial literacy and decision support. Accordingly, this study proposes to conduct a clinical trial literacy intervention using AI-powered chatbots among haematological malignancy patients. Through a randomised controlled trial (RCT), it aims to evaluate the impact of AI-assisted health education on patients' understanding of clinical trials and intention to participate. This research seeks to validate the application value of AI technology in health education and explore scalable AI-assisted health education intervention models.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of artificial intelligence technology in health education, focusing on haematological cancer patients' awareness of and intention to participate in clinical trials. Through an AI-robot-mediated clinical trial science communication intervention, the research will systematically assess its impact on patients' cognitive levels, attitudes, and participation intentions, exploring a scalable new model for AI-assisted health interventions.

Specific objectives include: (1) Investigating current levels of clinical trial awareness and participation attitudes among haematological malignancy patients; (2) Assessing the practical impact of AI-bot-delivered clinical trial awareness interventions on patients' understanding and intention to participate; (3) Exploring the feasibility and scalability of AI-assisted health education in promoting patient engagement in clinical trials.

ELIGIBILITY:
Inclusion Criteria (1) Aged ≥18 years with clear consciousness; (2) Diagnosed with haematological malignancy meeting clinical treatment criteria (WHO criteria); (3) Capable of understanding health education content and possessing basic communication skills; (4) Willing to participate in this study and sign an informed consent form.

Exclusion Criteria

(1) Patients with concomitant cognitive impairment, psychiatric disorders, or other conditions severely affecting comprehension; (2) Anticipated hospital stay of less than 3 days, rendering completion of the intervention unfeasible; (3) End-of-life palliative care; (4) Previous participation in other clinical trial education programmes.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2025-06-28 (Actual); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
intention to participate | The first day of patient enrolment and the seventh day following completion of the one-week intervention
  Measurement via a questionnaire on patients' intention to participate in clinical trials and influencing factors.

SECONDARY OUTCOMES:
User experience | The seventh day following completion of the one-week intervention
  Through questionnaires on intention to use and satisfaction with robots, alongside interview guidelines, we gathered patients' willingness to use intelligent robots and their satisfaction, perceptions, and feedback regarding the robots' role in supporting health education.

CONTACTS AND LOCATIONS:
Overall Officials: Fuling Fu Zhou, Study Director — Zhongnan Hospital of Wuhan Universty
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No